CLINICAL TRIAL: NCT04546282
Title: Mechanisms of Resistance to 3rd Generation Thyrosine Kinase Inhibitors in Lung Cancer
Brief Title: Resistance to Oral Therapy in Lung Cancer
Acronym: RESTKI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0519
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: 3rd Tyrosine kinase inhibitor; Cell free DNA; Mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — cell free DNA extracted from blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osimertinib treated patients: Patients with metastatic adenocarcinoma of the lung for whom a 3rd generation TKI therapy is proposed and a search for resistance mutation by blood analysis as part of the usual management.
  Interventions: Other: Description of the molecular alterations detected in blood samples of patients treated by osimertinib

INTERVENTIONS:
Other: Description of the molecular alterations detected in blood samples of patients treated by osimertinib — Description of the molecular alterations detected in blood samples of patients treated by osimertinib. This test is usualyy performed routinely to detect conventional mutations including EGFR T790M. We performed panel of genes screeining based on next generation sequencing. Thius, iIn some cases, new mutations can be detected by this assay.

SUMMARY:
In the management of non-small cell lung cancer of the adenocarcinoma type, different therapeutic strategies can be proposed. These strategies are defined according to the results of a biological analysis of blood and/or tissue samples from the lung tumor. Mutations in the tumor DNA are sought. Thus, patients with sensitizing mutations can benefit from a treatment with a 3rd generation tyroine kinase inhibitor (TKI) whose efficacy has been widely demonstrated. Patients without tumor mutations will not benefit. However, resistance to TKIs appears after a certain time, often linked to the appearance of new mutations in the tumor. For this reason, blood biologic analyses are regularly performed to search for the emergence of resistance mutations and to propose a therapeutic alternative as soon as possible.

These analyses are performed routinely in the laboratory. In the course of these analyses, the investigators have identified conventional mutations but also new mutations not previously described in the literature.

Our objective is to list all the molecular abnormalities revealed during blood biological analyses, to determine their frequency and to study whether certain abnormalities can be linked to resistance to TKI.

ELIGIBILITY:
Inclusion Criteria:

* advanced non-small cell lung cancer stage IIIB/IV
* Documentation of activating EGFR mutations (exon 19 deletions or exon 21 L858R substitution mutations) at the time of initial diagnosis
* Patient may receive up to one line of third EGFR TKI
* Plasma sample testing performed to detect EGFR TKI resistance

Exclusion Criteria:

* Patients have other concurrent cancers
* Patients who are not eligible receive TKI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-11-28 (Actual)

PRIMARY OUTCOMES:
Description of the molecular alterations detected in patients treated with 3rd TKI and assessment link with progression free survival and overall survival features. | The analysis of the TKI effectiveness and the appearance of mutations will be performed over a period of 24 months.
  This retrospective study will collate the molecular alterations detected during routine analysis. The elements extracted from the file will be age, sex, type of tumor and clinical-histological characteristics, dates of diagnosis and start of treatment. In addition, information on the dates of appearance of resistances (radiographic or clinical) will also be provided.
  No additional analysis will be performed since the study will consist of the analysis of data generated by the analyses performed in the context of patient management and biological monitoring.
  This research does not aim to modify your care. There will be no additional consultation or examination, nor will there be any changes in the treatment prescribed by your doctor.

SECONDARY OUTCOMES:
Frequency of detected molecular alterations | The analysis of the TKI effectiveness and the appearance of mutations will be performed over a period of 24 months.
  Frequency of detected molecular alterations

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Solassol, Study Director — UH Montpellier
Locations (1):
- University Hospital, Montpellier, Hérault, France